CLINICAL TRIAL: NCT07295977
Title: The Effect of Dehydration on Natural Dental Fluorescence: A Clinical Evaluation
Brief Title: Effect of Dehydration on Dental Fluorescence
Status: Active, not recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MUDHF-2025-83
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Evaluate the Fluorescence of Natural Tooth Following Dehydration
Keywords: fluorescence; dehydration; teeth
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: Dehydration of teeth will be assessed at baseline, at the 5th minute, and at the 10th minute using three different evaluation techniques.
  Interventions: Diagnostic Test: Digital photograph with Ashur plaque indicator; Diagnostic Test: Digital photographs with the Led lights (365 nm); Diagnostic Test: The QLF (Quantitative Light-Induced Fluorescence- 405 nm) images

INTERVENTIONS:
Diagnostic Test: Digital photograph with Ashur plaque indicator — Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Ashur plaque indicator (405 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the Ashur device (1/125, f/22, ISO 25600). To ensure standardization all images will be captured in a dark room.
Diagnostic Test: Digital photographs with the Led lights (365 nm) — Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Led lights (365 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the LED lights (1/125, f/22, ISO 8000). To ensure standardization, the LED lights will be stabilized on the flash brackets at a 45° angle on both sides, and all images will be captured in a dark room.
Diagnostic Test: The QLF (Quantitative Light-Induced Fluorescence- 405 nm) images — The images obtained using the QLF (Quantitative Light-Induced Fluorescence- 405 nm) device will be recorded. QLF images will be obtained with its own camera.

SUMMARY:
A cheek retractor will be placed to ensure consistent isolation throughout the procedure. Dehydration will be assessed at baseline, at the 5th minute, and at the 10th minute using three different evaluation techniques. At each time point, digital photographs will be captured under two distinct fluorescence light sources to document changes visually. In addition, fluorescence images will be obtained using the QLF (Quantitative Light-Induced Fluorescence) device to provide objective, quantitative data. All images will be recorded and analyzed digitally to evaluate dehydration-related changes in fluorescence. The aim of our study is to clinically evaluate the changes in the fluorescence properties of natural tooth following dehydration.

DETAILED DESCRIPTION:
According to the power analysis, the required number of teeth was 69, with 95% statistical power and a 5% alpha error level. The study will be conducted at the Clinic of the Department of Restorative Dentistry, Marmara University Faculty of Dentistry. Individuals with caries-free teeth, no enamel defects, no restorations on tooth surfaces, no visible plaque, and adequate cognitive ability to read and understand the informed consent form will be included in the study. Those with teeth exhibiting discoloration or with systemic conditions or medication use that may cause structural changes on the tooth surfaces will be excluded. Maxillary and mandibular anterior teeth will be evaluated.

A cheek retractor will be placed in the patients' mouths, and baseline, 5th-minute, and 10th-minute dehydration will be evaluated using three different techniques. Digital photographs will be taken at baseline and post-procedure under two different fluorescence light sources (Ashur plaque indicator (405 nm), and Led lights (365 nm)), and the images obtained using the QLF (Quantitative Light-Induced Fluorescence- 405 nm) device will be recorded. Analyses will be carried out digitally. Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the LED lights (1/125, f/22, ISO 8000) and for the Ashur device (1/125, f/22, ISO 25600). To ensure standardization, the LED lights will be stabilized on the flash brackets at a 45° angle on both sides, and all images will be captured in a dark room. QLF images will be obtained with its own camera. The photographs and the QLF images will be analyzed using Adobe Photoshop software, and color changes will be determined based on ∆E values. For each method ∆E values will be calculated individually, there will be 3 different ∆E values (baseline and 5th-minute, baseline and 10th-minute, 5th-minute and 10th-minute). For ∆E calculations, the CIEDE2000 formula will be used, employing the measured L*, a*, b* and L*, c*, h* values obtained from baseline, 5th-minute and 10th-minute images. For the digital measurements, the intraobserver variability will be assessed, and after obtaining a high level of agreement, the study will be initiated. In statistical analyses, normality will be assessed using the Shapiro-Wilk test; repeated-measures ANOVA will be used if normal distribution is present, and the Friedman test will be applied if normality is not observed. A significance level of p<0.05 will be accepted.

The aim of this clinical study is to clinically evaluate the changes in the fluorescence properties of natural teeth following dehydration.

The hypotheses of the study (H1) are as follows:

1. The change in the fluorescence properties of natural teeth after dehydration exceeds clinically acceptable thresholds.
2. There is a significant difference among the various fluorescence evaluation methods used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with caries-free teeth, no enamel defects, no restorations on tooth surfaces, no visible plaque, and adequate cognitive ability to read and understand the informed consent form.

Exclusion Criteria:

* Individuals with teeth exhibiting discoloration or with systemic conditions or medication use that may cause structural changes on the tooth surfaces.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with caries-free teeth, no enamel defects, no restorations on tooth surfaces, no visible plaque, and adequate cognitive ability to read and understand the informed consent form will be included in the study. Those with teeth exhibiting discoloration or with systemic conditions or medication use that may cause structural changes on the tooth surfaces will be excluded. Maxillary and mandibular anterior teeth will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Digital photograph with Ashur plaque indicator | baseline
  Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Ashur plaque indicator (405 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the Ashur device (1/125, f/22, ISO 25600). To ensure standardization all images will be captured in a dark room.
Digital photographs with the Led lights (365 nm) | baseline
  Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Led lights (365 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the LED lights (1/125, f/22, ISO 8000). To ensure standardization, the LED lights will be stabilized on the flash brackets at a 45° angle on both sides, and all images will be captured in a dark room.
The QLF (Quantitative Light-Induced Fluorescence- 405 nm) images | baseline
  The images obtained using the QLF (Quantitative Light-Induced Fluorescence- 405 nm) device will be recorded. QLF images will be obtained with its own camera. All images will be captured in a dark room.
Digital photograph with Ashur plaque indicator | at 5th minute
  Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Ashur plaque indicator (405 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the Ashur device (1/125, f/22, ISO 25600). To ensure standardization all images will be captured in a dark room.
Digital photographs with the Led lights (365 nm) | at 5th minute
  Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Led lights (365 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the LED lights (1/125, f/22, ISO 8000). To ensure standardization, the LED lights will be stabilized on the flash brackets at a 45° angle on both sides, and all images will be captured in a dark room.
The QLF (Quantitative Light-Induced Fluorescence- 405 nm) images | at 5th minute
  The images obtained using the QLF (Quantitative Light-Induced Fluorescence- 405 nm) device will be recorded. QLF images will be obtained with its own camera. All images will be captured in a dark room.
Digital photograph with Ashur plaque indicator | at 10th minute
  Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Ashur plaque indicator (405 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the Ashur device (1/125, f/22, ISO 25600). To ensure standardization all images will be captured in a dark room.
Digital photographs with the Led lights (365 nm) | at 10th minute
  Digital photographs will be taken at baseline and post-procedure under the fluorescence light source (Led lights (365 nm). Images will be captured with a Sony Alpha 7iii (Sony, Japan) digital camera equipped with a 90-mm macro lens. Camera settings will be adjusted for the LED lights (1/125, f/22, ISO 8000). To ensure standardization, the LED lights will be stabilized on the flash brackets at a 45° angle on both sides, and all images will be captured in a dark room.
The QLF (Quantitative Light-Induced Fluorescence- 405 nm) images | at 10th minute
  The images obtained using the QLF (Quantitative Light-Induced Fluorescence- 405 nm) device will be recorded. QLF images will be obtained with its own camera. All images will be captured in a dark room.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared after the publication of the study
Supporting Information: Study Protocol, SAP, ICF, CSR